CLINICAL TRIAL: NCT01619891
Title: VitamIN D Treating patIents With Chronic heArT failurE
Acronym: VINDICATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, KK Witte, Senior Lecturer in Cardiology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR/J00281X/1
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D 100mcg per day
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Standard optimal therapy
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 100mcg per day

SUMMARY:
Despite recent advances and even when receiving optimal therapy, patients with chronic heart failure (CHF) suffer poor quality of life, with recurrent hospitalisations and persistent symptoms. The investigators have shown that patients attending the Leeds Integrated Heart Failure Service are also frequently deficient in vitamin D and that the severity of the deficiency relates to the levels of symptoms, exercise capacity, diuretic requirements and response to optimal medical therapy. Vitamin D contributes to cardiac and skeletal muscle contractile function, immune function, pancreatic insulin release, and neuro-hormonal homeostasis. A randomised, placebo-controlled proof of concept study in 60 CHF patients has demonstrated improvements in submaximal exercise capacity and symptoms. VINDICATE will be a randomised, placebo-controlled developmental clinical study in 250 patients with CHF and vitamin D deficiency. The present study is designed to detect whether vitamin D has pathophysiologically important effects, as well as providing preliminary evidence of efficacy and safety by examining cardiac function (using cardiac magnetic resonance imaging) and submaximal exercise capacity (by 6-minute walk test). This will provide pertinent data to inform a larger multi-centre efficacy and effectiveness study.

DETAILED DESCRIPTION:
This is a randomized placebo-controlled trial of vitamin D versus placebo in people with heart failure. Primary endpoint is 6 minute walk distance.

ELIGIBILITY:
Inclusion Criteria:

* Class II or III CHF
* Stable symptoms (on otherwise optimally tolerated medical therapy)
* Able to give written informed consent

Exclusion Criteria:

* Currently taking vitamin D supplementation
* Untreated valvular heart disease
* Existing class I indication for vitamin D therapy
* History of primary hyperparathyroidism, tuberculosis, sarcoidosis, malignancy or hypercalcaemia
* Heart failure due to anaemia or thyrotoxicosis
* Renal failure (GFR <30l/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
6 minute walk distance | After one year

SECONDARY OUTCOMES:
Left ventricular function by Cardiac Magnetic Resonance | At one year
Peak exercise capacity | At one year
Biochemical changes | At one year (but also throughout)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus K Witte, MD, Principal Investigator — University of Leeds
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Witte KK, Byrom R, Gierula J, Paton MF, Jamil HA, Lowry JE, Gillott RG, Barnes SA, Chumun H, Kearney LC, Greenwood JP, Plein S, Law GR, Pavitt S, Barth JH, Cubbon RM, Kearney MT. Effects of Vitamin D on Cardiac Function in Patients With Chronic HF: The VINDICATE Study. J Am Coll Cardiol. 2016 Jun 7;67(22):2593-603. doi: 10.1016/j.jacc.2016.03.508. Epub 2016 Apr 4. PMID 27058906